CLINICAL TRIAL: NCT02103036
Title: Valuation of the Low Back Pain Treated With Different Types of Active Exercises in Women
Acronym: ECOLUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Rovira i Virgili (Other)
Collaborators: Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Principal Investigator, M. Rosa Nogués, Pharm. D., University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECOLUM
Record Dates: First submitted 2014-03-19; First posted 2014-04-03 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Core stability exercise; Back school; TENS; Infra- red light
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core Stability Exercises (Experimental): Core Stability Exercises:
  20 sessions, distributed daily, from Monday to Friday. The first 5 sessions are common in all patients in the study, and involves the application of infrared light (IR) (10 minutes) and TENS (20 minutes) to treat acute pain. From session number 6 to session 20, the patients will receive IR + TENS 2 days a week, and the other 3 days IR+TENS+Core Stability Exercises (25-30 minutes).
  Interventions: Procedure: Core Stability Exercises (CSE); Device: TENS; Device: Infra-red
- Traditional Back School (Experimental): Traditional Back School:
  20 sessions, distributed daily, from Monday to Friday. The first 5 sessions are common in all patients in the study, and involves the application of infrared light (IR) (10 minutes) and TENS (20 minutes) to treat acute pain. From session number 6 to session 20, the patients will receive IR + TENS 2 days a week, and the other 3 days IR+TENS+Traditional Back School (25-30 minutes).
  Interventions: Procedure: Traditional Back School; Device: TENS; Device: Infra-red

INTERVENTIONS:
Procedure: Core Stability Exercises (CSE) — The increase in intra-abdominal pressure stiffens and strengthens the relevant structural support around the spine, compacts the arthrogenic structures and in combination with abdominal contraction, it can encourage a rigid cylinder and stiffness to occur around the spine. The relevant anatomy in these type of exercises are deep muscles like transversus abdominous, multifidus or pelvic floor. The participants will have to do 10 different exercises. They will have to perform from 8 to 10 repetitions of every exercise, guided by a physical therapist. They will be recommended about making some series more at home, three days a week, when the treatment was finished.
  Other Names: Motor control exercises; Specific spinal stabilitation exercises
  Arms: Core Stability Exercises
Procedure: Traditional Back School — The back school exercises are based in the traditional activity used for improve the back pain symptoms using the breathing with the stretching of the trunk muscles, the erector spinae reinforcement, the abdominal reinforcement or the postural movements. The participants will have to do 10 different exercises. They will have to perform from 8 to 10 repetitions of every exercise, guided by a physical therapist. They will be recommended about making some series more at home, three days a week, when the treatment was finished.
  Arms: Traditional Back School
Device: TENS — Used equipment: MEGASONIC 313 P4 (Carin). Application program number 15: analgesic TENS with stimulation of afferent fibers.
  Type of current: two-phase TNS. Width of the impulse: 70µs. Frequency of the impulse: 100Hz. Train: Not. Pause / pause activates: Not. Time of treatment: 20 minutes.
  Other Names: Transcutaneous Electrical Nerve Stimulation
Device: Infra-red — Used equipment: INFRA - 2000 (Enraf Nonius) with the following parameters: 230 V / 50-60 Hz / 1.2 A
  Other Names: Infrared light

SUMMARY:
The purpose of the study is determine whether the Core Stability Exercise is more effective than the traditional Back School for low back pain (LBP) in women.

DETAILED DESCRIPTION:
The aim of this study is to check what kind of exercises are the best to treat LBP with regard to clinical improvements. The secondary objectives are: to determine which treatment is more effective in improving pain in the fewest sessions possible, to determine the involvement of inflammatory biomarkers in the development of pain and revalue the results after one month of having finishing treatment.

The project is a longitudinal, single-blind and randomized study with two treatment groups:

GROUP 1: Infrared light+ Transcutaneous Electrical Nerve Stimulation (TENS) + Core Stability Exercises.

GROUP 2: Infrared light + Transcutaneous Electrical Nerve Stimulation (TENS) + Traditional Back School.

Duration of treatment: 4 weeks. The participants will performe the exercises in 20 daily sessions (Monday to Friday) guided by a physiotherapist. Following treatment with the physiotherapist, the participants should perform the exercises at home for 4 weeks at a rate of three times per week.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 70 years.
* Diagnosis of back pain from a trauma.
* Untreated pain (except acetaminophen).
* Informed consent.

Exclusion Criteria:

* Algic process in the lumbar spine of infectious, neoplastic, metastasis, osteoporosis, inflammatory arthritis or fractures.
* Cognitive impairment of any etiology.
* Exercise intolerance for any reason.
* Patients who have completed physical therapy in the last 3 months.
* Patients who have received infiltration injections in the last 6 weeks.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Visual Scale Analogue (VAS) | Pain was measured at the beginning of the study (session 0), and changes are evaluated again at sessions 10, 20, and 1 month later.
  The VAS scale represents the pain intensity on a line of 10 cm, and one end there are the words "no pain" and the other end "the worst imaginable pain" written the distance in centimetres from the "no pain" point to the place marked by the patient represents the intensity of pain.

SECONDARY OUTCOMES:
Changes in the Roland- Morris Disability Questionnaire | Disability was measured at the beginning of the study (session 0), and changes are evaluated again at sessions 10, 20, and 1 month later.
  It consists of 24 items, which reflect limitation in different activities of daily living attributed by the patient to LBP. The patient must mark each item that applies to her current status. Scoring is also simple and fast; each checked item receives a score of 1, so scores range between 0 (no disability caused by LBP) and 24 (the maximum possible disability).

OTHER OUTCOMES:
Questionnaire of Physical Activity (ClassAF) | The physical activity will be measured at the beginning of the study (session 0).
  Is a method developed by the Health Department of the Catalan Government. The ClassAF is a comprehensive questionnaire which contains a few items (1-4) to measure the general level of Physical Activity, it is calculated in METS (basal metabolic expenditure: mlO2/kg.min) and it allows to classify people into physically active or physically inactive.
Changes in the biomarkers: Tumor Necrosis Factor (TNF-Alpha) and Interleukin 10 (IL-10) | The concentrations of these biomarkers will be measured at the beginning (session 0) and changes will be evaluated again at the end of the treatment (session 20).
  These two cytokines are parameters to indicate the inflammation levels. Their concentrations are measured using commercial ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Nogués, Pharm.D., Study Director — Faculty of Medicine and Health Sciences. Rovira i Virgili University. Spain.
Locations (1):
- Faculty of Medicine and Health Sciences, Reus, Tarragona, Spain

REFERENCES:
- [Derived] Minobes-Molina E, Nogues MR, Giralt M, Casajuana C, de Souza DLB, Jerez-Roig J, Romeu M. Effectiveness of specific stabilization exercise compared with traditional trunk exercise in women with non-specific low back pain: a pilot randomized controlled trial. PeerJ. 2020 Nov 27;8:e10304. doi: 10.7717/peerj.10304. eCollection 2020. PMID 33312766